CLINICAL TRIAL: NCT05171699
Title: Effect of Electroacupuncture in Patients With Sepsis Associated Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Director, Tianjin Nankai Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NKYY-EA-SAE
Record Dates: First submitted 2021-10-13; First posted 2021-12-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Electroacupuncture; Sepsis; Sepsis-associated Brain Injury
MeSH Terms: conditions — Sepsis | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture (Experimental): The investigators choose Zusanli (ST36) and Baihui (DU20) acupoints to investigate the effect of electroacupuncture on patients with sepsis-associated brain injury.
  Interventions: Other: electroacupuncture
- shame electroacupuncture (Sham Comparator): The shame electroacupuncture were performed at a shallow depth and 1 mm lateral to Zusanli (ST36) and Baihui (DU20) acupoints.
  Interventions: Other: shame electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — The patients in Group EA received electroacupuncture at Zusanli (ST36) (located 5 mm below the head of the inferior fibula and 2 mm lateral to the anterior tibial tuberosity) and Baihui (DU20) (located in the midpoint of the parietal bone) acupoints, the stainless steel acupuncture needles were connected to a Hans acupoint nerve stimulator and inserted into the acupoints.
  Arms: electroacupuncture
Other: shame electroacupuncture — The patients in Group SEA received electroacupuncture at a shallow depth and 1 mm lateral to Zusanli (ST36) (located 5 mm below the head of the inferior fibula and 2 mm lateral to the anterior tibial tuberosity) and Baihui (DU20) (located in the midpoint of the parietal bone) acupoints, the stainless steel acupuncture needles were connected to a Hans acupoint nerve stimulator and inserted into the acupoints.
  Arms: shame electroacupuncture

SUMMARY:
To investigate the effect of electroacupuncture on patients with sepsis-associated brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age is between 20 and 80 years.
2. Patients meeting the diagnosis of sepsis-associated brain injury.
3. Patients who agreed to accept this trial and signed the informed consent form.

Exclusion Criteria:

1. Patients with a history of brain injury, stroke, epilepsy, cognitive impairment, or mental illness prior to admission.
2. Patients who were also involved in any other interventional study.
3. Due to hearing or vision loss, or any other situation that may seriously interfere with study data collection.
4. Patients who refused to participate in this study.
5. The pregnancy test was positive or is currently breastfeeding.
6. Any other situation that the investigator believed might be detrimental to participant in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
neuron specific enolase,NSE | Change of NSE from Baseline at 7 days
  Serum index of sepsis-associated brain injury.
sTREM2 | Change of sTREM2 from Baseline at 7 days
  Serum index of sepsis-associated brain injury.
soluble protein-100β,S100β | Change of S100β from Baseline at 7 days
  Serum index of sepsis-associated brain injury.

SECONDARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation，APACHE II | Change of APACHE II from Baseline at 7 days
  To assess the severity of the disease.
Glasgow Coma Scale，GCS | Change of GCS from Baseline at 7 days
  To assess the degree of coma.
Montreal Cognitive Assessment (MoCA) scale | Change of MoCA from Baseline at 7 days
  Rapid screening for cognitive function abnormalities。

OTHER OUTCOMES:
length of stay in hospital | 2 months
fatality rate at 28 days after discharge | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Nankai Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No